CLINICAL TRIAL: NCT05682716
Title: Application of Intraoperative Transesophageal Echocardiography Imaging of Vein and Controlled Low Central Venous Pressure in Early Prediction and Intervention of Acute Renal Injury Associated With Cardiac Surgery
Brief Title: Application of Intraoperative Transesophageal Echocardiography Imaging of Vein and CLCVP in Early Prediction and Intervention CSA-AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT20230104
Record Dates: First submitted 2023-01-04; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Acute Kidney Disease; Postoperative complications of cardiac surgery; Transesophageal echocardiography
MeSH Terms: conditions — Acute Kidney Injury | interventions — Technology; Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Controlled low central venous pressure (CLCVP) technology
  Interventions: Combination Product: Controlled low central venous pressure (CLCVP) technology; Drug: Nitroglycerin
- control group (No Intervention)

INTERVENTIONS:
Combination Product: Controlled low central venous pressure (CLCVP) technology — Controlled low central venous pressure (CLCVP) technology: after cardiopulmonary bypass, pumping nitroglycerin (0.2-1 ug/kg * min) and other methods until the end of surgery to maintain the central venous pressure below 10 mmHg.
  Arms: Intervention group
Drug: Nitroglycerin — nitroglycerin (0.2-1 ug/kg * min)
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn about in postoperative acute kidney injury in cardiac surgery. The main questions it aims to answer are:

* Intraoperative Transesophageal Ultrasound Doppler venous imaging can be used to predict the occurrence of cardiac surgery associated acute kidney injury (CSA-AKI ) in the early stage by observing the changes of renal vein, portal vein and hepatic vein blood flow patterns, calculating the renal vein stasis index and portal vein pulsatility index, and evaluating the degree of venous congestion.
* Controlled low central venous pressure (CLCVP) technology can reduce the occurrence of CSA-AKI by reducing venous congestion and increasing renal perfusion pressure.

Participants will receive Transesophageal Ultrasound Doppler during cardiac surgery. If the participant is assigned to the intervention group, if the central venous pressure of the participant is ≥ 10mmHg 30 minutes after the end of cardiopulmonary bypass, he will receive nitroglycerin pumped to apply the controlled low central venous pressure (CLCVP) technology; If participants are assigned to the control group, no intervention measures will be taken.

The researchers will compare the intervention group with the control group to see the occurrence of AKI and AKD after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients aged above 18 years undergoing coronary artery bypass graft or heart valve surgery under cardiopulmonary bypass.

Exclusion Criteria:

1. Patients with CKD history, end-stage renal disease and renal transplantation before operation
2. Used nephrotoxic drugs within two weeks before operation
3. Known Renal Artery Stenosis and Renal Malformations
4. There are contraindications for transesophageal ultrasound Doppler evaluation of esophageal space occupying lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Level of Serum creatinine | Before operation to 90 days after operation
  SCR

SECONDARY OUTCOMES:
Neutrophil gelatinase associated lipid transporter (NGAL) | Before operation to 2 hours after operation
  Neutrophil gelatinase associated lipid transporter
Kidney Injury Molecule-1 (KIM-1) | Before operation to 12 hours after operation
  Kidney Injury Molecule-1

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen L, Hong L, Ma A, Chen Y, Xiao Y, Jiang F, Huang R, Zhang C, Bu X, Ge Y, Zhou J. Intraoperative venous congestion rather than hypotension is associated with acute adverse kidney events after cardiac surgery: a retrospective cohort study. Br J Anaesth. 2022 May;128(5):785-795. doi: 10.1016/j.bja.2022.01.032. Epub 2022 Mar 4. PMID 35249707
- [Result] Lopez MG, Shotwell MS, Morse J, Liang Y, Wanderer JP, Absi TS, Balsara KR, Levack MM, Shah AS, Hernandez A, Billings FT 4th. Intraoperative venous congestion and acute kidney injury in cardiac surgery: an observational cohort study. Br J Anaesth. 2021 Mar;126(3):599-607. doi: 10.1016/j.bja.2020.12.028. Epub 2021 Feb 4. PMID 33549321